CLINICAL TRIAL: NCT06840730
Title: Investigation of the Relationship Between Clinical Results of Onabotulinum Toxin a Application and Pain Mediators in the Treatment of Myospasm-Related Masticatory Muscle Disorder
Brief Title: Efficiency of Botulinum Toxin Type-a in the Management of the Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Salih Eren Meral, DDS phd, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-23004
Record Dates: First submitted 2025-02-13; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Myofascial Pain - Dysfunction Syndrome of TMJ
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- botulinum toxin (Experimental): TX-A will be injected into the masseter and temporalis muscles (30 and 15 units per side, respectively) following a standardized protocol.
  Interventions: Drug: Botulinum Toxin A (Botox )

INTERVENTIONS:
Drug: Botulinum Toxin A (Botox ) — TX-A will be injected into the masseter and temporalis muscles (30 and 15 units per side, respectively) following a standardized protocol.

SUMMARY:
**Study Title:** Investigation of the Relationship Between Clinical Outcomes and Pain Mediators in the Treatment of Masticatory Muscle Disorders Associated with Myospasm Using Onabotulinum Toxin A

**Study Importance:** Temporomandibular disorders (TMD) are a major cause of chronic orofacial pain, affecting 5-12% of the population. Masticatory muscle disorders (MMD) are a common subgroup of TMD, ranging from localized myalgia to fibromyalgia. Myospasm is characterized by sudden pain, malocclusion, and limited jaw movement, while myalgia includes localized, myofascial, and referred pain patterns. The etiology of MMD is complex, involving neuromuscular dysfunction, inflammation, and increased acetylcholine activity at the neuromuscular junction. Various mediators, including CGRP, substance P, and inflammatory cytokines, play a role in sensitization and pain perception.

**Objective:** This study aims to evaluate the effectiveness of onabotulinum toxin A (BTX-A) in patients with MMD who have not responded to conventional non-invasive treatments. It hypothesizes that BTX-A reduces pain by decreasing inflammatory cytokines and neuropeptides associated with pain.

**Methodology:**

* **Study Design:** Prospective observational clinical study.
* **Participants:** Patients diagnosed with MMD based on RDC/TMD criteria, who have not improved with conventional treatments.
* **Exclusion Criteria:** Conditions such as pregnancy, metabolic disorders, trauma, systemic diseases, and medication use that could interfere with results.
* **Intervention:** BTX-A will be injected into the masseter and temporalis muscles (30 and 15 units per side, respectively) following a standardized protocol.
* **Data Collection:**
* Before (T0) and one month after (T1) treatment.
* Clinical assessments include maximum mouth opening (MMO), pain levels (VAS), and oral health impact profile (OHIP-14).
* Blood and saliva samples will be analyzed for IL-1, IL-6, TNF-α, CGRP, and NGF using ELISA.
* **Statistical Analysis:** Dependent t-test or Wilcoxon signed-rank test will be used to compare pre- and post-treatment values. Correlations between biomarker levels and pain reduction will be analyzed using Spearman correlation.

**Expected Outcomes:**

* Significant reduction in pain and improvement in MMO.
* Decreased levels of inflammatory and neuropeptide biomarkers.
* Evaluation of saliva as a non-invasive medium for biomarker analysis, potentially guiding future diagnostic and monitoring strategies.

**Significance:** This study provides insights into the pathophysiology of MMD and the efficacy of BTX-A in pain management, potentially offering an alternative therapeutic approach for patients resistant to conventional treatments.

ELIGIBILITY:
Inclusion Criteria: Patients diagnosed with MMD based on RDC/TMD criteria, who have not improved with conventional treatments.

-

Exclusion Criteria:Conditions such as pregnancy, metabolic disorders, trauma, systemic diseases, and medication use that could interfere with results

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Significant reduction in pain and improvement in mouth openins. | 1 month
  Significant reduction in pain and improvement in maximum mouth openings in post-operative measurements.

SECONDARY OUTCOMES:
Evaluation of the levels of inflammatory and neuropeptide biomarkers in serum and saliva specimens. | 1 month
  Serum and salivary levels of inflammatory and neuropeptide biomarkers, including nerve growth factor, calcitonin gene-related peptide, and interleukin 1 beta tumor necrosis factor-alpha, in serum specimens will be evaluated on the post operative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided